CLINICAL TRIAL: NCT07369596
Title: Impact of Chemotherapy Dose Reductions on Survival Outcomes Among Older NSCLC Patients Without Actionable Mutations: A Retrospective Cohort Study.
Brief Title: Impact of Chemotherapy Dose Reductions on Survival Outcomes Among Older NSCLC Patients Without Actionable Mutations
Status: Recruiting | Type: Observational
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Poh Mau Ern, Professor Dr, University of Malaya
Other Study IDs: 20258615434
Record Dates: First submitted 2025-12-22; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Carcinoma NSCLC
Keywords: NSCLC; older patients; chemotherapy
MeSH Terms: interventions — Progression-Free Survival

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal dose group: Patients receiving standard dose of chemotherapy
  Interventions: Other: Progression free survival; Other: Overall survival
- Dose reduction group: Patients receiving lower doses of chemotherapy
  Interventions: Other: Progression free survival; Other: Overall survival

INTERVENTIONS:
Other: Progression free survival — PFS
Other: Overall survival — OS

SUMMARY:
Evidence suggests that appropriately selected older adults can tolerate standard-dose chemotherapy and achieve survival outcomes comparable to younger patients. However, older adults are usually under-represented in clinical trials and often receive reduced doses of chemotherapy due to concerns regarding age-related frailty, polypharmacy, and toxicity.

This study seeks to evaluate chemotherapy dosing patterns and associated survival outcomes in older patients.

DETAILED DESCRIPTION:
Lung cancer remains the leading cause of cancer-related mortality globally, responsible for approximately 1.8 million deaths annually. Non-small cell lung cancer (NSCLC) comprises about 85% of all lung cancer cases, with adenocarcinoma (ADC) now the predominant histological subtype. In Malaysia, NSCLC is similarly the most common form of lung cancer, with high proportions of EGFR and ALK mutations in certain subgroups.

Despite the emergence of targeted therapy and immunotherapy, cytotoxic chemotherapy, particularly platinum-based doublets remains the backbone of treatment for many NSCLC patients lacking actionable mutations. These patients often present with advanced disease and limited survival prospects, with median overall survival (OS) of 8- 10 months. These includes older patients with advanced NSCLC and no actionable mutations who depend on chemotherapy for disease control.

Clinical decisions regarding dosing are frequently influenced by perceptions of frailty rather than individual fitness. Evidence suggests that appropriately selected older adults can tolerate standard-dose chemotherapy and achieve survival outcomes comparable to younger patients. However, older adults are usually under-represented in clinical trials and often receive reduced doses of chemotherapy due to concerns regarding age-related frailty, polypharmacy, and toxicity. This raises an important question: does dose reduction compromise survival outcomes in older NSCLC patients?

This study seeks to address this knowledge gap by retrospectively evaluating chemotherapy dosing patterns and associated survival outcomes in older patients treated at three centres in Malaysia: Universiti Malaya Medical Centre (UMMC), Hospital Tengku Ampuan Afzan, Kuantan and Hospital Wanita dan Kanak-kanak, Likas, Sabah and one centre in Hong Kong: Queen Mary Hospital, The University of Hong Kong. It will evaluate whether chemotherapy dose reductions are associated with poorer survival outcomes in older NSCLC patients. It will also assess clinical predictors such as ECOG performance status, BMI, comorbidities, and gender to identify factors influencing treatment tolerance and survival.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years
* Histologically confirmed stage IV NSCLC
* Negative for EGFR mutation, ALK rearrangement, and ROS1 fusion
* Treated with at least ONE cycle of first-line chemotherapy

Exclusion Criteria:

* Patients who received targeted therapy or immunotherapy as monotherapy in the first-line setting
* Incomplete survival data

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Retrospective cohort study using data from three centres in Malaysia from 2020 to 2025. All patients aged ≥65 years with advanced/metastatic NSCLC and no actionable driver mutations who received AT LEAST ONE CYCLE of first-line chemotherapy will be included in the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To compare the overall survival (OS) between older NSCLC patients treated with standard-dose versus reduced-dose first-line platinum-doublet chemotherapy OR single agent non-platinum chemotherapy. | From enrollment to the end of study on 31 Dec 2026

SECONDARY OUTCOMES:
To compare the progression free survival (PFS) between older NSCLC patients treated with standard-dose versus reduced-dose first-line platinum-doublet chemotherapy OR single agent non-platinum chemotherapy. | From enrollment to end of study on 31 Dec 2026
To assess objective response rates in patients who complete FOUR cycles of chemotherapy. | From enrollment to end of study period on 31 Dec 2026

CONTACTS AND LOCATIONS:
Overall Officials: Mau Ern Poh, MBBS, Principal Investigator — Universiti Malaya
Locations (4):
- Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong
- Malaysia (3):
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - Hospital Wanita dan Kanak-Kanak Sabah, Kota Kinabalu, Sabah
  - Universiti Malaya Medical Centre, Kuala Lumpur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 10. Tan DSW, Yom SS, Tsao MS, et al. The international association for the study of lung cancer consensus statement on optimizing management of EGFR mutation-positive non-small cell lung cancer: Status in 2016. Journal of Thoracic Oncology 2016; 11, 946-963.
- [Background] 9. Solomon BJ, Mok T, Kim DW, et al. First-line crizotinib versus chemotherapy in ALK-positive lung cancer. New England Journal of Medicine 2014; 371, 2167-2177.
- [Background] 8. Mok TS, Wu YL, Thongprasert S, et al. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. New England Journal of Medicine 2009; 361, 947-957.
- [Background] 7. Sedrak MS, Sun CL, Liu X, et al. Aging and tolerance to chemotherapy: Impact of dose reduction and treatment delays on survival outcomes. Journal of Clinical Oncology, 2021 39, 1714-1723.
- [Background] 6. Hurria A, Kris MG, and Hudis C. Management of lung cancer in older adults. CA: A Cancer Journal for Clinicians 2003; 53, 325-341.
- [Background] 5. Maione P, Perrone F, Gallo C, et al. Pretreatment quality of life and functional status assessment significantly predict survival of elderly patients with advanced non-small cell lung cancer receiving chemotherapy: A prognostic analysis of the Multicenter Italian Lung Cancer in the Elderly Study. Journal of Clinical Oncology 2005, 23, 6865-6872.
- [Background] 4. Sundararajan V., Hershman DL, Grann VR, Jacobson JS, and Neugut, AI. Variations in the use of chemotherapy for elderly patients with advanced ovarian cancer: a population-based study. Gynecologic Oncology 2018, 115, 344-350
- [Background] 3. Liam, Chong-Kin, Toh-Yoon Evelyn Goh, Nur Syafikah Shamsudin, and Chee-Chee Khoo. 2022. "Driver Gene Alterations and PD-L1 Expression in Non-Small Cell Lung Cancer and Their Association with Smoking and Gender in a Malaysian Population." Asian Pacific Journal of Cancer Prevention 23 (6): 1911-1917.
- [Background] 2. Hurria A, Togawa K., Mohile SG, Owusu C, Klepin HD, et al. Predicting chemotherapy toxicity in older adults with cancer: a prospective multicenter study. Journal of Clinical Oncology 2011, 29, 3457-3465.
- [Background] 1. Hamaker ME., Schiphorst AHW, ten Bokkel Huinink D, Schaar C, & van Munster BC. The effect of a geriatric evaluation on treatment decisions for older cancer patients-a systematic review. Acta Oncologica 2014, 53, 289-296.